CLINICAL TRIAL: NCT01485159
Title: Airflow Limitation in Cardiac Diseases in Europe
Acronym: ALICE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115398
Record Dates: First submitted 2011-11-17; First posted 2011-12-05 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: prevalence; COPD; emphysema; co-morbidities; ischemic heart disease; chronic bronchitis; spirometry; burden
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Myocardial Ischemia; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — In patients that specifically consent, blood samples will be taken for future analysis of the genetic links between COPD and cardiovascular disease
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: All subjects enrolled in the study
  Interventions: Procedure: Spirometry

INTERVENTIONS:
Procedure: Spirometry — assessment of lung function by spirometry

SUMMARY:
This is a cross-sectional, observational study, investigating the point prevalence of Airflow Limitation in current or former smokers with established ischemic heart disease. The study will recruit up to 3000 patients from cardiology clinics at hospitals across Europe.

DETAILED DESCRIPTION:
Airflow limitation (AL) occurs in a number of respiratory diseases including asthma and COPD; in middle-aged and older patients it typically represents Chronic Obstructive Pulmonary Disease (COPD), and is associated with a high degree of co-morbidity which includes cardiovascular diseases (CVD) and risk factors such as hypertension and diabetes.

COPD often goes undiagnosed, especially in patients with established coronary disease because COPD and cardiovascular diseases share a major etiological factor: smoking.

This cross-sectional, observational study, investigating the prevalence of AL in current or former smokers with established ischemic heart disease, aims increase the knowledge and understanding of COPD in this patient population, and to highlight the burden of comorbid disease in these patient

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥40 years;
* Current or former smokers with ≥10 pack years;
* Subjects attending outpatient cardiac clinic (or equivalent) fulfilling any of the following criteria:

  1. Documented history of an Ischemic event,
  2. Current diagnosis of stable IHD (including history of acute Myocardial Infarction (MI) and angina pectoris) as diagnosed in accordance with ESC guidelines
  3. Receiving regular therapy for IHD for >1yr, Subjects meeting these criteria will be eligible for the study, even if they have other cardiac diseases or other co-morbidities;
* Subjects willing and able to sign study consent form.

Exclusion Criteria:

* Subjects for whom spirometry is contraindicated;
* Subjects with recent surgery or MI (within 1 month); lower respiratory tract infection or pneumothorax (within 2 months); or stroke (within 12 months);
* Subjects with a pre-existing condition which, in the opinion of the investigator, would compromise the safety of the subject in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending outpatient cardiology clinics with a history of Ischemic Heart Disease
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of Airflow Limitation | 1 day
  Prevalence of AL as defined by Forced Expired Volume in 1 second (FEV1)/Forced Volume Capacity (FVC) < 0.70 (post bronchodilator)

SECONDARY OUTCOMES:
Severity of AL | 1 day
  Severity of AL as determined by predicted FEV1 (post-bronchodilator) - mild: ≥80%, moderate: 50-80%, severe: 30-50%, very severe: <30%, or <50% plus chronic respiratory failure
prevalence of restrictive AL | 1 day
  Prevlence of restrictive AL FEV1/FVC ≥0.70 and a predicted FVC <80% (pre bronchodilator)
Prevalence of AL | 1 day
  Prevalence of AL as defined by FEV1 below the lower limit of normal
Presence of past history of AL/COPD | 1 day
  prevalence of documented evidence of COPD, chronic bronchitis or emphysema
COPD Assessment test™ (CAT) | 1 day
  Health status questionnaire on burden of airflow limitation (CAT)
Short Form 12 (SF12) | 1 day
  General health status questionnaire (SF12)
Cardiac Health Profile (CHP) | 1 day
  Health status questionnaire on burden of cardiac disease
Healthcare resource utilisation | within previous 12 months
  Number of emergency room visits and hopsital admissions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- GSK Investigational Site, Ghent, Belgium
- GSK Investigational Site, Toulouse, France
- Germany (2):
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Thessaloniki, Greece
- GSK Investigational Site, Dublin, Ireland
- Italy (2):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Tradate (VA), Lombardy
- Netherlands (2):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Sneek
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
- Sweden (2):
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Malmo

REFERENCES:
- [Derived] Franssen FM, Soriano JB, Roche N, Bloomfield PH, Brusselle G, Fabbri LM, Garcia-Rio F, Kearney MT, Kwon N, Lundback B, Rabe KF, Raillard A, Muellerova H, Cockcroft JR. Lung Function Abnormalities in Smokers with Ischemic Heart Disease. Am J Respir Crit Care Med. 2016 Sep 1;194(5):568-76. doi: 10.1164/rccm.201512-2480OC. PMID 27442601